CLINICAL TRIAL: NCT05466669
Title: Prediction of Post-TIPS Hepatic Encephalopathy in Patients With Liver Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Christian Labenz, Priv.-Doz. Dr. med., Johannes Gutenberg University Mainz
Other Study IDs: 20221
Record Dates: First submitted 2022-07-13; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Hepatic Encephalopathy; Liver Cirrhosis
Keywords: Liver Cirrhosis; Hepatic Encephalopathy; Transjugular Intrahepatic Portosystemic Shunt; TIPS; Post-TIPS Hepatic Encephalopathy; Post-TIPS HE; Minimal Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood (EDTA, serum). Portal vein blood (EDTA, serum). Hepatic vein blood (EDTA, serum).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prediction of hepatic encephalopathy after insertion of a transjugular intrahepatic portosystemic stent shunt (post-TIPS HE) are critical for patient selection prior to TIPS insertion, and a currently unmet, clinically highly relevant need. In this prospective multicenter observational cohort study, the investigators aim to evaluate the ability of Stroop EncephalApp and the simplified Animal Naming Test (S-ANT1) in comparison to the goldstandard PHES to predict the occurence of post-TIPS HE in patients with decompensated liver cirrhosis. Moreover, secondary aims of this study include the detection of potential blood based biomarkers for prediction of post-TIPS HE and the predictive value of frailty and quality of life/sleep prior to TIPS insertion.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis (clinical, sonographic, CT-morphological, laparoscopic or histological)
* TIPS indication: refractory ascites or secondary prophylaxis after variceal bleeding
* Age ≥ 18 years
* Ability to give consent
* Consent to the study after comprehensive information

Exclusion Criteria:

* Contraindication against TIPS insertion
* Lack of consent
* History of liver transplantation
* Preemptive TIPS
* Emergency TIPS
* Severe neurological comorbidities

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants are recruited from the outpatient clinic or from the regular wards of the hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2025-02-10 (Estimated); Study Completion 2025-02-10 (Estimated)

PRIMARY OUTCOMES:
Prediction of post-TIPS HE using established tests | 12 months
  Evaluation of the predictive value of S-ANT1 and Stroop EncephalApp compared with PHES (gold standard) for predicting post-TIPS HE within the first 12 months after TIPS implantation.

SECONDARY OUTCOMES:
Evaluation of candidate inflammatory biomarkers (using the Olink target 96 panel) for predicting of post-TIPS HE | 12 months
  Evaluation of exploratory candidate inflammatory biomarkers derived from peripheral blood and analyzed using the validated Olink target 96 panel for the prediction ofpost-TIPS HE.
Evaluation of the impact of frailty, assessed by the Liver Frailty Index (LFI) on the risk of post-TIPS HE. | 12 months
  The presence of frailty - using the validated LFI - will be assessed in each patient prior to TIPS implantation and 1, 3 and 6 months after TIPS implantation. The full range of the LFI is 1.0-7.0 (with a higher score indicating that the patient is more frail)
Longitudinal assessment of health-related quality of life using the Chronic Liver Disease Questionnaire (CLDQ) | 12 months
  Health-related quality will be assessed in each participant using the validated CLDQ. Quality of life will be assessed at baseline and 1-, 3- and 6- months post-TIPS implantation.
Longitudinal assessment of cognitive function after TIPS insertion | 12 months
  Assessment of longitudinal changes in PHES, Stroop EncephalApp and S-ANT1 after TIPS implantation. The tests will be applied to all patients at baseline and at 1-, 3- and 6- months post-TIPS implantation.
Evaluation of serum Neurofilament Light Chains (sNfL) and Glial fibrillary acidic protein (GFAP) for predicting of post-TIPS HE | 12 months
  Evaluation of the usefulness of sNfL and GFAP for predicting post-TIPS HE during follow-up. sNfL and GFAP will be determined from blood obtained prior to TIPS implantation using a single molecule array (SiMoA technology).
Longitudinal assessment of sleep quality using the Pittsburgh Sleep Quality Index (PSQI) | 12 months
  Sleep quality will be assessed in each participant using the validated PSQI. Sleep quality will be assessed at baseline and 1-, 3- and 6- months post-TIPS implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Labenz, MD, Principal Investigator — Department of Internal Medicine I, University Medical Center of the Johannes Gutenberg-University Mainz
Locations (2):
- Germany (2):
  - Department of Internal Medicine I, University Medical Center of the Johannes Gutenberg-University Mainz, Mainz, Rhineland-Palatinate
  - Department of Medicine I, University Hospital Schleswig-Holstein, Lübeck, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kabelitz MA, Gairing SJ, Tiede A, Schleicher EM, Ahl LG, Wagner L, Zucker-Reimann F, Rieland H, Mauz JB, Weinmann-Menke J, Meyer BC, Pitton MB, Wedemeyer H, Galle PR, Sandmann L, Maasoumy B, Labenz C. Impact of Frailty on the Prognosis of Patients With Liver Cirrhosis Undergoing Insertion of a TIPS. Aliment Pharmacol Ther. 2026 Jan;63(1):109-118. doi: 10.1111/apt.70315. Epub 2025 Aug 1. PMID 40751304